CLINICAL TRIAL: NCT06067074
Title: Is it Cost-effective With Volar Plating Surgery Compared to Non-operative Treatment for Distal Radius Fracture in the Elderly?
Brief Title: Cost-effectiveness, Volar Locking Plate or Non-operative Treatment Distal Radius Fracture
Acronym: HE-VOCAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Cecilia Mellstrand Navarro, associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: study2
Record Dates: First submitted 2022-05-12; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Radius Fractures; Aged; Cost-Benefit Analysis; Wrist Fracture; Quality of Life; Wrist Injuries; Postoperative Complications; Health Care Utilization
MeSH Terms: conditions — Radius Fractures; Wrist Fractures; Wrist Injuries; Postoperative Complications; Patient Acceptance of Health Care | interventions — Casts, Surgical

STUDY DESIGN:
Intervention Model Description: Parallell study arms with the intervention volar locking plate and control treatment forearm cast. We investigate the difference in health cost between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volar Locking Plate (Experimental): Surgery with a Volar Locking Plate due to displaced distal radius fracture
  Interventions: Procedure: Volar Locking Plate
- Non-operative treatment group (Experimental): Patients allocated to non-operative treatment received a plaster cast for 4-5 weeks.
  Interventions: Procedure: Plaster Cast

INTERVENTIONS:
Procedure: Volar Locking Plate — Surgery
  Arms: Volar Locking Plate
Procedure: Plaster Cast — Non-operative treatment with a plaster cast
  Arms: Non-operative treatment group

SUMMARY:
A cost-utility analysis based on an earlier published RCT comparing surgery with volar locking plate to non-operative treatment for the elderly with a displaced distal radius fracture.

DETAILED DESCRIPTION:
Study design: A cost-utility analysis of a patient population included in a previous published randomized controlled trial.

Patient population:140 patients 70 years of age or older with a displaced distal radius fracture that met the inclusion and no exclusion criteria at Danderyd Hospital or Södersjukhuset Hospital were randomized to volar locking plate or non-operative treatment with a cast.

Primary outcome: Incremental cost-effectiveness ratio (ICER) at 1 and 3 years.

Data collection: Prospectively collected clinical data is available for 4, 12, weeks, 1 and 3 years. Costs will be analysed regarding surgical equipment, inpatient stay, surgical time. Prescriptions of analgesics and antibiotics as well as inpatient and outpatient consumption over a three years period after the injury will be retrieved from the Swedish National Board of Health and Welfare.The life expectancy adjusted life years (QALYs) is calculated from prospectively collected results from EQ-5D.

ELIGIBILITY:
Inclusion Criteria

* patient >70 years
* wrist radiograph >20° dorsal tilt and/or +/-4 mm axial shortening

Exclusion Criteria

* Former disability of either wrist
* Intra-articular fractures with a step-off of >1 mm or a gap of > 1 mm (at Sodersjukhuset Hospital)
* High-energy trauma (Sodersjukhuset Hospital)
* Associated ulnar fracture
* Injury to ipsilateral upper extremity
* Rheumatoid arthritis or other severe joint disorders
* Dementia or Pfeiffer score of <5 at Sodersjukhuset Hospital and <8 at Danderyd Hospital
* Drug or alcohol abuse or psychiatric disorder
* Dependency in activities of daily living
* Patient not a resident within the catchment area of the 2 centers
* Fracture diagnosed >3 days from injury at Sodersjukhuset Hospital and >6 days at Danderyd Hospital
* Patient not fit for surgery or American Society of Anesthesiologists class 4

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-11-04 (Estimated); Study Completion 2024-11-04 (Estimated)

PRIMARY OUTCOMES:
Incremental Cost-Effectiveness Ratio (ICER) at 1 year. | 1 year
  difference in cost divided by difference in quality of life

SECONDARY OUTCOMES:
Absolute cost difference | 1 and 3 years
  difference in cost between treatments
ICER at 3 years | 3 years
  difference in cost divided by difference in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Olof Sköldenberg, professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Department of Clinical Sciences, Danderyd Hospital, Division ot Ortopeadics, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No